CLINICAL TRIAL: NCT02701361
Title: Mobile Mindfulness to Improve Psychological Distress After Critical Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Washington (Other); University of Pennsylvania (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00064250; R34AT008819 (NIH)
Record Dates: First submitted 2016-02-24; First posted 2016-03-08 (Estimated); Results first posted 2018-01-10 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Psychological Distress; Depression; Anxiety; Post-traumatic Stress Disorder; Informal Caregivers; Family Members
Keywords: mindfulness; critical illness; intensive care unit; mindfulness-based stress reduction
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Critical Illness | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Education group (Active Comparator): A care condition in which an educational program relevant to critical illness is presented in a web-based format similar to the other arms. Telephone calls will be used to answer questions and assist with web content.
  Interventions: Behavioral: education
- Standard mindfulness (Experimental): Receives audiovisual mindfulness content via internet plus 1 call per week from a trained mindfulness expert.
  Interventions: Behavioral: standard mindfulness
- Mobile mindfulness (Experimental): Receives audiovisual mindfulness content via web-app. Will receive at least 1 call from a trained mindfulness expert, though up to 4 total calls based on symptoms / request.
  Interventions: Behavioral: mobile mindfulness

INTERVENTIONS:
Behavioral: mobile mindfulness — Receives audiovisual mindfulness content via internet plus call depending on symptoms or request.
  Arms: Mobile mindfulness
Behavioral: standard mindfulness — Receives weekly calls from mindfulness expert for 4 weeks.
  Arms: Standard mindfulness
Behavioral: education — Receives web-based content about critical illness topics. Also receives two calls from study team to describe materials and answer questions about materials.
  Arms: Education group

SUMMARY:
Many survivors of the intensive care unit (ICU) suffer from persistent symptoms of depression, anxiety, and post-traumatic stress disorder (PTSD). In this study, the investigators will test the impact of mindfulness to address this distress.

DETAILED DESCRIPTION:
A majority of the >1 million people who require life support in an intensive care unit (ICU) now survive. As survival has improved however, growing numbers suffer not only from subsequent physical disability, but also persistent symptoms of depression, anxiety, and post-traumatic stress disorder (PTSD). Few interventions address ICU survivors' psychological distress. Fewer still address the physical, geographical, and logistical barriers to receiving post-discharge support that medically ill populations encounter. Consequently, this population suffers with an unmet need of great public health importance.

Mindfulness is an adaptable self-regulation practice that alleviates psychological distress symptoms using a variety of meditative techniques, typically taught face-to face over months. As an extension of standard mindfulness practices, the investigators developed a telephone-/web-delivered mobile mindfulness-based training (mMBT) system informed by ICU survivors' input that could address medically ill patients' delivery barriers. The investigators' recent pilot study demonstrated early support for mMBT's feasibility and acceptability, now with enhanced content and electronic patient-reported outcomes capability.

The investigators' early work on mMBT, while promising, identified key knowledge gaps in population targeting, plausible ranges of psychological distress estimates relevant to study design, and assurance of acceptability that must be addressed before a definitive clinical trial is conducted. Therefore, the study team proposes a 2-year pilot study in which 90 ICU survivors are randomized to an education control, 'standard' telephone sessions of mMBT, or self-directed / app-based mMBT. A mixed methods approach will be used to determine treatment effect.

ELIGIBILITY:
Inclusion Criteria (the investigators will target patients at high risk for psychological distress):

* age ≥18 years
* acute cardiorespiratory failure managed in an intensive care unit
* reside at home before hospital admission (i.e., not in a facility)

  * Respiratory failure, ≥1 of these:
* mechanical ventilation via endotracheal tube for ≥ 12 hours
* non-invasive ventilation (CPAP, BiPAP) for > 4 hours in a 24 hour period provided for acute respiratory failure in an ICU (not for obstructive sleep apnea or other stable use)
* high flow nasal cannula or face mask O2 with FiO2 ≥ 0.5 for ≥4 hours

  * Cardiac / circulatory failure, ≥1 of these:
* use of vasopressors for shock of any etiology for > 1 hour
* use of inotropes for shock of any etiology for > 1 hour
* use of aortic balloon pump for cardiogenic shock

Exclusion Criteria (present before consent): Patients will be excluded if they have characteristics that would prohibit adequate participation including:

* pre-existing significant cognitive impairment (e.g., dementia)
* treated for severe or unstable mental illness within 6 months preceding current admission (e.g., depression with psychosis, suicidality, schizophrenia as per medical record)
* hospital inpatient within 3 months before current admission
* active substance abuse at the time of admission
* lack of decisional capacity [*'Decisional capacity' is defined as the ability to participate in effective decision making and provide informed consent. That is, in the judgment of the examiner, the patient, after reading the IRB approved patient consent document (or having it read to them) can (a) generally understand the terms of participation in the study: the purpose of the study, what will be required of study participants; the potential risks, benefits and alternatives of study participation; pros & cons of study involvement and (b) can communicate a choice in his/her own words (or write on a communication board)]
* current significant cognitive impairment (≥3 errors on the Callahan cognitive status screen; see below)
* need for a translator because of poor English fluency [many study instruments are not validated in other languages]
* expected survival <6 months per attending physician
* ICU length of stay >30 days
* lack of either:
* reliable or sufficient smartphone with cellular data plan or
* reliable computer online access plus telephone access
* unable to complete study procedures as determined by study staff
* discharge to a location other than a home setting
* complex medical care expected soon after discharge (e.g., multiple planned surgeries, transplantation evaluation (including outpatient daily cardiopulmonary rehabilitation), extensive travel needs for hemodialysis, disruptive chemotherapy or XRT regimen, etc)

Other issues relevant to the consent process:

* unable to approach patient for logistical reasons (e.g., off ward in test at time of approach, etc)
* patient discharged before consent could be obtained
* patient dies before consent obtained

Patient exclusion criteria present after consent but before randomization:

After providing informed consent, patients will become ineligible if any of the following are present:

* they become too ill to participate (or die)
* they exhibit significant cognitive disability
* they exhibit suicidality
* patient was unexpectedly discharged to location other than a home setting and then did not arrive home within 1 month from hospital discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E Cox, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University, Durham, North Carolina
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cox CE, Porter LS, Buck PJ, Hoffa M, Jones D, Walton B, Hough CL, Greeson JM. Development and preliminary evaluation of a telephone-based mindfulness training intervention for survivors of critical illness. Ann Am Thorac Soc. 2014 Feb;11(2):173-81. doi: 10.1513/AnnalsATS.201308-283OC. PMID 24303911
- [Derived] Cox CE, Hough CL, Jones DM, Ungar A, Reagan W, Key MD, Gremore T, Olsen MK, Sanders L, Greeson JM, Porter LS. Effects of mindfulness training programmes delivered by a self-directed mobile app and by telephone compared with an education programme for survivors of critical illness: a pilot randomised clinical trial. Thorax. 2019 Jan;74(1):33-42. doi: 10.1136/thoraxjnl-2017-211264. Epub 2018 May 23. PMID 29793970

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 90 participants signed consent; 2 participants who signed consent were later found not to be eligible(88 eligible). 80 participants were randomized
Period: Overall Study
Arm/Group | Mobile Mindfulness | Standard Mindfulness | Education Group
Started | 31 | 31 | 18
Completed | 22 | 28 | 16
Not Completed | 9 | 3 | 2
Not completed — Lost to Follow-up | 5 | 2 | 1
Not completed — Withdrawal by Subject | 4 | 0 | 0
Not completed — timed out in rehab center | 0 | 1 | 0
Not completed — incarceration | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Mindfulness | Standard Mindfulness | Education Group | Total
Number analyzed (Participants) | 31 | 31 | 18 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (15.3) | 48.1 (16.1) | 53.3 (12.6) | 49.5 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 8 | 35
  Male | 19 | 16 | 10 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 31 | 30 | 18 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2 | 4
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 3
  Black or African American | 4 | 9 | 5 | 18
  White | 23 | 20 | 10 | 53
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent of Eligible Participants Who Provided Consent
Description: Percent of eligible participants who provided consent. Because this includes eligible yet not-as-yet randomized participants, there are no study arm differences analyzed. This is a feasibility measure. Target is 70%.
Time Frame: pre-randomization
Population: 121, not 90 subjects, are analyzed because this outcome measure applies to a pre-consent and pre-randomization time period.
Measure: Count of Participants; unit: Participants
Groups:
- All Eligible Subjects Approached to Participate in the Study: All eligible subjects approached to participate in the study.
Arm/Group | All Eligible Subjects Approached to Participate in the Study
Number analyzed (Participants) | 121
Participants | 90

2. Primary Outcome: Percent of Eligible Participants Who Provide Informed Consent and Were Randomized
Description: Percent of eligible participants who provide informed consent and were randomized. A measure of feasibility. Target is 60%.
Time Frame: randomization
Population: Following consent, two participants were found to be ineligible.
Measure: Count of Participants; unit: Participants
Groups:
- All Eligible Participants: All eligible participants.
Arm/Group | All Eligible Participants
Number analyzed (Participants) | 88
Participants | 80

3. Primary Outcome: Client Satisfaction Questionnaire (CSQ) Score
Description: Acceptability was measured with the adapted Client Satisfaction Questionnaire (CSQ), which assesses credibility and satisfaction (range 9 [low, a worse outcome] to 36 [highest, a better outcome]). Target is mean score >10.
Time Frame: 1 month post-randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mobile Mindfulness | Standard Mindfulness | Education Group
Number analyzed (Participants) | 22 | 28 | 16
units on a scale | 27.6 (3.8) | 29.4 (3.3) | 25.7 (3.2)

4. Primary Outcome: System Usability Scale (SUS)
Description: Usability of the mobile app was assessed with open-ended participant feedback and with the 10-item System Usability Scale (SUS; 0 [lowest] to 100 [highest]). A SUS score above a 68 would be considered above average and anything below 68 is below average.
Time Frame: 1 month post-randomization
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Mobile Mindfulness
Number analyzed (Participants) | 22
units on a scale | 86.5 (13.3)

5. Primary Outcome: Percent of Randomized Participants Who Drop Out of Study
Description: A feasibility measure. Target is 20% or less.
Time Frame: baseline, end of study (approx. 4 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Mindfulness | Standard Mindfulness | Education Group
Number analyzed (Participants) | 31 | 31 | 18
Participants
  before intervention initiated | 7 | 2 | 0
  after intervention initiated | 2 | 1 | 2

6. Primary Outcome: Percent of Participants Who Have Neither Dropped Out Nor Died Who Complete Telephone Interviews
Description: Percent of participants who have neither dropped out nor died who complete telephone interviews. A feasibility measure. Target is 75%.
Time Frame: baseline, end of study (approx. 4 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Mindfulness | Standard Mindfulness | Education Group
Number analyzed (Participants) | 22 | 28 | 16
Participants | 22 | 28 | 16

7. Primary Outcome: Percent of Participants in the Self-directed MBT Group Who Complete Weekly Surveys
Description: A feasibility measure. Target is 60%. Note that this is for completion of ALL FOUR weekly surveys.
Time Frame: baseline, end of study (approx. 4 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Mindfulness
Number analyzed (Participants) | 22
Participants | 17

8. Primary Outcome: Percentage of Self-directed MBT Sessions Attended by Eligible Participants
Description: A feasibility measure. Target is 50% among those who neither dropped out nor died.
Time Frame: baseline, end of study (approx. 4 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Mindfulness
Number analyzed (Participants) | 22
Participants | 22

9. Primary Outcome: Visual Analog Satisfaction Scale
Description: A measure of acceptability of the intervention. Target mean score is 75% or greater.
Time Frame: after intervention completion, up to 8 weeks post-randomization
Population: measure was mistakenly omitted from study CRF and therefore data not collected.
Arm/Group | Mobile Mindfulness
Number analyzed (Participants) | 0

10. Primary Outcome: Number of Participant Clicks on Study Website
Description: A usability measure obtained using Google Analytics.
Time Frame: baseline, end of study (approx. 4 months)
Measure: Mean (Standard Deviation); unit: clicks
Arm/Group | Mobile Mindfulness
Number analyzed (Participants) | 22
clicks | 188.4 (220.8)

11. Secondary Outcome: Change in Psychological Distress Symptoms as Measured by the Patient Health Questionnaire (PHQ) Scale
Description: Depression symptoms were assessed with the PHQ-9, a 9-item scale (range 0 [no distress] to 27 [high distress]); symptom severity is interpreted as mild (5-9), moderate (10-14), moderately severe (15-19), and severe (20-27).
Time Frame: Between randomization and 3 months post-randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mobile Mindfulness | Standard Mindfulness | Education Group
Number analyzed (Participants) | 31 | 31 | 18
units on a scale | -4.8 [-6.6 to -2.9] | -3.9 [-5.6 to -2.2] | -3.0 [-5.3 to -0.8]

12. Secondary Outcome: Change in Distress Associated With Physical Symptoms
Description: The PHQ-10 (Patient Health Questionnaire) was used to measure distress associated with physical symptoms (range 0 [none] to 30 [very troublesome]).
Time Frame: Between randomization and 3 months post-randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mobile Mindfulness | Standard Mindfulness | Education Group
Number analyzed (Participants) | 31 | 31 | 18
units on a scale | -5.3 [-7.0 to -3.7] | -3.7 [-5.2 to -2.2] | -4.8 [-6.8 to -2.7]

13. Secondary Outcome: Change in Mindfulness Skills
Description: Mindfulness skills were measured with the Cognitive and Affective Mindfulness Scale-Revised (CAMS-R), a 12-item measure of mindful qualities (range 12 [low ability] to 48 [highest ability]).
Time Frame: Between randomization and 3 months post-randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mobile Mindfulness | Standard Mindfulness | Education Group
Number analyzed (Participants) | 31 | 31 | 18
units on a scale | 0.7 [-1.7 to 3.0] | -0.9 [-3.1 to 1.3] | -1.3 [-4.1 to 1.5]

14. Secondary Outcome: Change in Psychological Distress Symptoms as Measured by the GAD-7
Description: Anxiety symptoms were measured using the Generalized Anxiety Disorder 7-item scale (GAD-7; range 0 [no distress] to 21 [high distress]); symptom severity is interpreted as mild (5-9), moderate (10-14), and severe (15-21).
Time Frame: Between randomization and 3 months post-randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mobile Mindfulness | Standard Mindfulness | Education Group
Number analyzed (Participants) | 31 | 31 | 18
units on a scale | -2.1 [-3.7 to -0.5] | -1.6 [-3.0 to -0.1] | -0.6 [-2.5 to 1.3]

15. Secondary Outcome: Change in Psychological Distress Symptoms as Measured by the PTSS
Description: The Post Traumatic Stress Scale (PTSS), a 10-item scale (range 10 [no symptoms] to 70 [high burden of symptoms]), was used to assess PTSD symptoms; >20 represents clinically important symptoms.
Time Frame: Between randomization and 3 months post-randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mobile Mindfulness | Standard Mindfulness | Education Group
Number analyzed (Participants) | 31 | 31 | 18
units on a scale | -2.6 [-6.3 to 1.2] | -2.2 [-5.6 to 1.2] | -3.5 [-8.0 to 1.0]

16. Secondary Outcome: Change in the Avoidance Domain of the Brief COPE Scale
Description: Coping skills were measured with the Brief COPE scale (range 10 [low use] to 40 [highest use]). The Brief COPE is a self-report questionnaire used to assess a number of different coping behaviors and thoughts a person may have in response to a specific situation.
Time Frame: Between randomization and 3 months post-randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mobile Mindfulness | Standard Mindfulness | Education Group
Number analyzed (Participants) | 31 | 31 | 18
units on a scale | -0.5 [-1.9 to 1.0] | 1.3 [-0.03 to 2.7] | -0.2 [-2.0 to 1.6]

17. Other Pre Specified Outcome: Usability Themes Developed From Semi-structured Participant Interviews
Description: A usability measure. Open-ended feedback questions will be arranged in themes.
Time Frame: end of study
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Mobile Mindfulness | Standard Mindfulness | Education Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/18
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2016-05-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT02701361/ICF_000.pdf
  • Study Protocol (2016-10-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT02701361/Prot_001.pdf
  • Statistical Analysis Plan (2016-05-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT02701361/SAP_003.pdf